CLINICAL TRIAL: NCT00225875
Title: Evaluation De l'Efficacité Du Rituximab (Mabthéra) Chez l'Adulte Atteint d'Un Purpura thrombopénique Auto-Immun Chronique Et sévère Et Candidat à La splénectomie
Brief Title: Study of the Effectiveness of Rituximab in Adults With Chronic and Severe Immune Thrombocytopenic Purpura and Candidate for a Splenectomy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Etablissement Français du Sang (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTAI
Record Dates: First submitted 2005-09-20; First posted 2005-09-26 (Estimated); Last update posted 2005-10-27 (Estimated); Status verified 2005-03

CONDITIONS: Autoimmune Thrombocytopenic Purpura
Keywords: Autoimmune thrombocytopenic purpura; Rituximab
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

INTERVENTIONS:
Drug: Mabthéra

SUMMARY:
The goal of this study is to evaluate the clinical effectiveness of the rituximab at the adults with a chronic immune thrombocytopenic purpura (>=6 months of evolution) and severe (platelets <= 30x109/L) and candidate to a splenectomy. The objective is to obtain after a treatment by the rituximab a satisfactory response to one year, defined by a number of platelets higher than 50x109/L and at least 2 times superior with the persistent initial figure without treatment during one year after the end of the treatment.

DETAILED DESCRIPTION:
Adults immune thrombocytopenic purpura has an evolution which is generally chronic defined by the persistence of the thrombocytopenia 6 months after the diagnosis. The treatment is then based on the splenectomy which is proposed by the majority of the teams when the platelets are lower than 30x109/L. The splenectomy is effective at 70 to 80 % of the patients whereas no medicamentous treatment makes it possible to obtain a comparable result. Nevertheless, it exposes to immediate post-operative complications and to a risk of mortal fulminant infections by encapsulated germs, in particular the pneumococcus. However, its long-term effectiveness is discussed with a risk of relapse which would reach 50 % for certain teams.

The rituximab could be an alternative to the splenectomy because of its great frequency of effectiveness and its good tolerance in the short and medium term. None the medicamentous treatments usually suggested in alternative to the splenectomy (disulone, danazol, immunosuppressors) indeed makes it possible to obtain an answer prolonged after the stop of therapeutic in a significant number of cases. Moreover, the use of the immunosuppressors such as the cyclophosphamide, the azathioprine or the ciclosporine appears contestable at this stage of the disease because of potential severity their side effects.The primary endpoint is satisfactory response to one year, defined by a figure of plates >=50x109/L and at least 2 times superior in the initial, and persistent figure without treatment during one year after the stop of the treatment by rituximab. Secondary objectives are incomplete response to one year, defined by a figure of platelets >= 30x109/L and < 50x109/L and at least twice the figure initial or > 50x109/L but lower than twice the persistent initial figure without treatment during one year after the end of the treatment by rituximab. Splenectomy at one year satisfactory Response to 2 years incomplete Response to 2 years Splenectomies at 2 years Tolerance of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Platelets <= 30x109/L in the absence of agglutinat
* Evolution of the PTAI >= 6 months starting from the date of the diagnosis
* Myélogramme normal and rich in mégacaryocytes
* Age >=18 years
* Among patients at which the treatments prescribed before (and in particular corticoids or intravenous immunoglobulins) did not have any effectiveness, even transitory, the diagnosis of ITP will have to be confirmed by an isotopic study of the 1/2 life of the plates.

Exclusion Criteria:

* Refusal of informed and enlightened assent written.
* Intermittent ITP defined by which has occurred of transitory periods of remissions variable length of the thrombocytopenia.
* Sick splenectomized whatever is the reason
* Splénomégalie
* Absence of vaccination against the pneumococcus
* Absence of vaccination against Haemophilus influenzae
* Previous of treatment by the rituximab
* Administration of a treatment known as active during the ITP other than corticoids in the 30 days which precede inclusion
* CIVD and/or weakens haemolytic with schizocytes
* Serology VIH or positive VHC, Ag positive HBs
* Rate of ALAT or ASAT higher than twice the higher limit of the normal of the laboratory
* Associated autoimmune anomalies:

  * Anti DNA and/or anti ECT (ENA) and/or anti Ro (SSA)
  * The presence isolated from antibody anti cores (nuclear anti factors) is not a criterion of exclusion.
  * Anticoagulant circulating of lupic type and/or antibody anticardiolipines with antecedent of thrombosis or spontaneous miscarriages with repetition (their isolated presence is not a criterion of exclusion)
  * Other autoimmune diseases: lupus (with at least 4 criteria of the ACR), polyarthrite chronic evolutionary, disease of Biermer, affected thyroid, weakens haemolytic autoimmune.
* Pregnant woman, breast feeding, woman in genital working life in the effective absence of contraception throughout treatment and 12 month after stop of the treatment.
* Evolutionary or previous cancer of malignant hemopathy
* Over-sensitiveness with murine proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2003-09; Study Completion 2007-07

PRIMARY OUTCOMES:
Satisfactory response to one year, platelets >=50x109/L and at least 2 times superior in the initial, and persistent figure without treatment during one year after the stop of the treatment.

SECONDARY OUTCOMES:
Incomplete response to one year,platelets >= 30x109/L and < 50x109/L and at least twice the figure initial or > 50x109/L but lower than twice the persistent initial figure without treatment during one year after the end of the treatment.
Splenectomy at one year satisfactory Response to 2 years Incomplete Response to 2 years Splenectomy at 2 years Tolerance of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Godeau, Professor, Principal Investigator — Henri Mondor University Hospital; Philippe Bierling, Professor, Principal Investigator — EFS
Locations (1):
- Hôpital Henri Mondor, Créteil, France

REFERENCES:
- [Background] Michel M, Chanet V, Galicier L, Ruivard M, Levy Y, Hermine O, Oksenhendler E, Schaeffer A, Bierling P, Godeau B. Autoimmune thrombocytopenic purpura and common variable immunodeficiency: analysis of 21 cases and review of the literature. Medicine (Baltimore). 2004 Jul;83(4):254-263. doi: 10.1097/01.md.0000133624.65946.40. PMID 15232313
- [Derived] Godeau B, Porcher R, Fain O, Lefrere F, Fenaux P, Cheze S, Vekhoff A, Chauveheid MP, Stirnemann J, Galicier L, Bourgeois E, Haiat S, Varet B, Leporrier M, Papo T, Khellaf M, Michel M, Bierling P. Rituximab efficacy and safety in adult splenectomy candidates with chronic immune thrombocytopenic purpura: results of a prospective multicenter phase 2 study. Blood. 2008 Aug 15;112(4):999-1004. doi: 10.1182/blood-2008-01-131029. Epub 2008 May 7. PMID 18463354